CLINICAL TRIAL: NCT01496677
Title: A Phase 1 Open-Label Study With Oral TR-701 Free Acid to Assess Pharmacokinetics, Safety, and Tolerability in Elderly Subjects
Brief Title: Pharmacokinetics, Safety, and Tolerability of TR-701 Free Acid (FA) in Elderly Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Trius Therapeutics LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1986-028; TR701-109 (Other: TriusRX Unique ID)
Record Dates: First submitted 2011-12-19; First posted 2011-12-21 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2017-10

CONDITIONS: Healthy Subjects
Keywords: volunteer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Elderly subjects (65 or older) (Experimental)
  Interventions: Drug: TR-701 FA 200 mg
- Younger adults (18-45 years old) (Experimental)
  Interventions: Drug: TR-701 FA 200 mg

INTERVENTIONS:
Drug: TR-701 FA 200 mg — Single oral tablet of TR-701 FA to elderly subjects
  Arms: Elderly subjects (65 or older)
Drug: TR-701 FA 200 mg — Single oral tablet of TR-701 FA to younger group (18-45 years old)
  Arms: Younger adults (18-45 years old)

SUMMARY:
To compare the pharmacokinetic (PK) profile of TR-700 in elderly subjects versus younger control subjects

DETAILED DESCRIPTION:
This is an open-label Phase 1 study of a single oral tablet of TR-701 FA 200 mg to compare the TR-700 PK profile in elderly subjects (age 65 years and older, with at least 5 subjects 75 years old or older) and younger control subjects (age 18 to 45 years).

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects in the following groups: An elderly subject at least 65 years of age. At least 5 subjects must be at least 75 years of age OR A matched-control subject between 18 and 45 years of age, inclusive
* BMI ≥18.0 kg/m2 and ≤35.0 kg/m2

Elderly Group

* Medical history, physical examination, and laboratory results consistent with stable health (as determined by the Investigator)

Control Group

* Medically stable with no clinically significant abnormalities

Exclusion Criteria:

* Significant, uncontrolled, or life-threatening condition or organ or system condition or disease (eg, impaired cognitive status, respiratory insufficiency, advanced malnutrition)
* Positive hepatitis B surface antigen, hepatitis C virus antibody, or human immunodeficiency virus antibody test result
* Previous inclusion in a TR-701 FA or TR-701 clinical study
* ECG finding of QTc interval >500 msec, or other clinically significant ECG abnormality at Screening
* Female subjects whom are pregnant, lactating or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2012-01-17 (Actual); Primary Completion 2012-02-28 (Actual); Study Completion 2012-02-28 (Actual)

PRIMARY OUTCOMES:
Compare PK profile of TR-700 FA in elderly subjects versus younger control subjects | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Philippe G Prokocimer, MD, Study Chair — Trius Therapeutics
Locations (1):
- Trius Investigator Site 001, Daytona Beach, Florida, United States

REFERENCES:
- [Derived] Flanagan SD, Minassian SL, Prokocimer P. Pharmacokinetics, Safety, and Tolerability of Tedizolid Phosphate in Elderly Subjects. Clin Pharmacol Drug Dev. 2018 Sep;7(7):788-794. doi: 10.1002/cpdd.426. Epub 2018 Jan 10. PMID 29319932